CLINICAL TRIAL: NCT04629820
Title: Effects of Near Vision Spectacle Correction on Work Productivity Among Textile Factory Workers in India
Brief Title: PROductivity Study of Presbyopia Elimination in Rural-dwellers II
Acronym: PROSPERII
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: VisionSpring (Other); University of Michigan (Other); Good Business Lab (Unknown); Zhongshan Ophthalmic Center, Sun Yat-sen University (Other); Clearly (Other)
Responsible Party: Principal Investigator, Nathan Congdon, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MHLS 20_82
Record Dates: First submitted 2020-10-21; First posted 2020-11-16 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Presbyopia
Keywords: Presbyopia; Refractive error; Work productivity; Spectacle wear compliance
MeSH Terms: conditions — Presbyopia; Refractive Errors | interventions — Eyeglasses

STUDY DESIGN:
Intervention Model Description: 800 textile workers aged 35 years and above with uncorrected presbyopia will be randomized to receive free glasses within one week of undergoing vision assessment, or free glasses at the end of the study assessment (3 months after vision assessment).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Study personnel assessing trial outcomes will be masked as to participants assignment, which will be simplified by the fact that there will be participants with and without glasses at both Intervention and Control. It is not ethical in this setting to provide Control participants with placebo treatment (glasses with zero power lenses), but participants will not be informed of either the overall design of the study or the explicit treatment intervention assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Workers assigned to the intervention group will receive free spectacles of a design they select, based on the worker's measured refractive power and dispensed one week later at the factory by the study ophthalmic personnel.
  Interventions: Device: Spectacles
- Control (No Intervention): Workers assigned to the Control group will receive similar free glasses at the end of the study assessment (3 months).

INTERVENTIONS:
Device: Spectacles — Intervention group workers receive free glasses within one week of undergoing vision assessment (September 2021). The assessment period will be three months
  Other Names: Near eyeglasses; Reading glasses
  Arms: Intervention

SUMMARY:
The investigators will conduct a randomized-controlled trial. The participants will be textile workers aged 35 years and above with uncorrected presbyopia who are employed by a single Indian garment manufacturer - employed by Shahi Exports Private Limited, Karnataka, India - at facilities equipped to measure individual productivity. PROSPER II will assess the impact of free reading glasses on productivity for workers in a textile factory.

DETAILED DESCRIPTION:
Globally, 3 billion people do not have the eyeglasses they need to earn, learn, travel safely in traffic and participate in civic life. Among these, 1.1 billion people lack a simple pair of reading glasses to correct impaired near vision, called presbyopia. Presbyopia, the essentially universal decline in unaided near vision that occurs with aging, is the world's most common cause of vision impairment. Loss of accommodation (ability to change focus from distance to near) due to presbyopia can begin as early as age 30 years, commonly becomes functionally apparent by 40, and is essentially complete by 55, meaning that presbyopia is most common at the height of the working years.

Study Plan: This is a randomized trial designed to assess the impact of free spectacles on workplace productivity among Indian textile workers.

Research question: Will providing free glasses to presbyopic Indian textile workers increase work productivity?

Design: Investigator-masked, multi-center randomized controlled trial

Rationale: Although presbyopia is safely, effectively and inexpensively treated with glasses, rates of optical correction in LMICs are as low as 10%. The global productivity loss due to uncorrected presbyopia has been estimated to exceed US$25 billion, and presbyopia is shown to be associated with significant impairment in activities of daily living. Few trials have been published which address the question of whether healthcare interventions can improve work performance as well as workplace retention, especially among persons over the age of 40 in low and middle-income countries (LMICs). The largest reported effect sizes among such trials was the PROSPER trial, which showed that providing inexpensive near vision glasses increased the daily weight of tea picked among presbyopic, mostly-female Indian agricultural workers by more than 5 kg (21.6%) compared to those in the control group. Costs were low, over half of pickers aged >= 40 years met criteria to receive glasses, and wearing compliance reached nearly 90%. There is interest to understand if these results from the agricultural setting can be extended to other financially-important sectors.

Methods : The investigators will enrol 800 textile workers aged 35 years and above with uncorrected presbyopia who are employed by Shahi Exports Private Limited in Karnataka, India. Eligible participants will be randomly assigned to Intervention and Control Groups (1:1). Intervention group participants will receive free reading glasses within a week of undergoing a vision screening at the factory. Control group participants will receive reading glasses at the end of the assessment period (three months after vision screening).

The main outcome 3 months later will be work productivity; secondary outcomes are change in skill grade, change in monthly wage, participants' adherence with spectacle wear, self-assessed self-efficacy score and change of quality of life scores. The intervention cost-effectiveness will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Aged 35 years and older
* Have presbyopia, defined as an unaided near visual acuity of N6.3 or worse in both eyes
* Require a new pair of glasses to improve their near vision
* Have a corrected near visual acuity of N4 or better in both eyes
* Have worked in Shahi's production department as tailors or Kajbutton operators for 6 weeks or more

Exclusion Criteria:

* Have ocular pathology in either eye detected during the eye examination, or history of such disease based on self-report
* Have a low likelihood of completing follow-up in the study due to current plans to move out of the area or leave employment at Shahi during the follow-up period

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Difference in change in mean efficiency between intervention and control group | Over the three month follow-up period from enrolment to study completion
  Efficiency is calculated as the proportion of target production realized by a worker per unit time

SECONDARY OUTCOMES:
Three-month change in skill grade | Between baseline and study end three months later
  Skill grade ranges from A triple star (highest) to A double star, A star, A, B, and C + (lowest)
Change in monthly wage | Between baseline and study end three months later
  Monthly wage (Factory administrative data)
Adherence with spectacle wear | Between baseline and study end three months later
  measured weekly by enumerator's unannounced observations of the presence of spectacles worn on the participant's face.
Group difference in three-month change in self-assessed self-efficacy scores | Between baseline and conclusion of the study three months later
  Self-assessed self-efficacy scores measured using the Cantril's Ladder, with the best possible score being a 10, and the worst being a 0 (Cantril's Ladder)
Group difference in three-month change of quality of life scores | Between baseline and conclusion of the study three months later
  Quality of life scores measured using the Andhra Pradesh Eye Disease Study (APEDS) Visual Function Questionnaire (VFQ), with a 5-point Likert scale: 1=No difficulty, 2=Little difficulty, 3=Moderate difficulty, 4=Great difficulty but still can manage, 5=Cannot manage. A highest score represents great difficulty in vision function. Minimum score = 16; Maximum score = 80.
Cost effectiveness | Between baseline and study end three months later
  Full programme costs per individual identified and corrected with presbyopia. Programme costs include costs incurred in screening test, glasses / replacement and direct/indirect costs for facilitating work-based site. Benefit will be measured using work productivity. We will report cost effectiveness distinguishing between study costs and program costs

CONTACTS AND LOCATIONS:
Overall Officials: Nathan G Congdon, MD, MPH, Principal Investigator — Queen's University, Belfast
Locations (1):
- Good Business Lab, Bengaluru, Karnataka, India

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available for download on the Queen's University Belfast website.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within 6 months of collection, for three years.
Access Criteria: Freely available
URL: http://qub.ac.uk

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-04-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT04629820/SAP_001.pdf